CLINICAL TRIAL: NCT05689463
Title: Evaluation of the Prevalence of BP180 and BP230 Autoantibodies in the Serum of Patients With Pruritus Under Immunotherapy
Acronym: BPA_immun
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/0429/HP
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Patients With Chronic Pruritus for More Than 1 Month Who Have Received Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with prurit (Experimental)
  Interventions: Biological: characterisation of immunoglobulin subclasses

INTERVENTIONS:
Biological: characterisation of immunoglobulin subclasses — For patients with positive anti BP180 and/or anti BP230 serology, a characterisation of the immunoglobulin subclasses will be performed

SUMMARY:
The aim of the study is to evaluate the prevalence of positive anti BP180 and/or anti BP230 serology in the serum of patients with chronic and diffuse pruritus for at least 1 month under immunotherapy and in the absence of obvious pruritic dermatosis (e.g. scabies, contact eczema...).

ELIGIBILITY:
Inclusion Criteria:

* Patient currently receiving immunotherapy (pembrolizumab, nivolumab, atezolizumab, durvalumab) as monotherapy or in combination OR patient who has received immunotherapy (pembrolizumab, nivolumab, atezolizumab, durvalumab) as monotherapy or in combination within the last 6 months.
* Patients with chronic (> 1 month) diffuse pruritus, which started after the start of immunotherapy and in the absence of an obvious pruritic dermatosis.
* Woman of childbearing age with effective contraception (see GTFG) (estrogen-progestin or intrauterine device or tubal ligation) for 1 month (negative urine/blood pregnancy test) or Postmenopausal woman: confirmatory diagnosis (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit)
* Major patient
* Patient having read and understood the information letter and signed the consent form
* Patient affiliated to a social security scheme

Exclusion Criteria:

Pruritus prior to immunotherapy. Bullous pemphigoid prior to immunotherapy End-stage chronic renal failure (GFR < 15ml/min or dialysis) Clinical jaundice or total bilirubin > 34 µmol/L Hepatic cholestasis Diabetes mellitus complicated by diabetic neuropathy. History of polycythemia vera History of Hodgkin's lymphoma iron deficiency anemia Current treatment including DPP-4 inhibitors (vildagliptin, linagliptin) Treatment with systemic corticosteroids or immunosuppressant for more than one month.

Pregnant or parturient or breastfeeding woman or absence of proven contraception

· Person deprived of liberty by an administrative or judicial decision or person placed under legal safeguard / sub-tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients on immunotherapy with chronic diffuse pruritus for at least 1 month with positive anti BP180 and/or anti BP230 serology | 1 day

SECONDARY OUTCOMES:
Number of anti-BP180 and/or anti-BP230 positive patients who will develop urticarial, eczematous or bullous disease | 30 days
Number of anti-BP180 and/or anti-BP230 positive patients who will develop urticarial, eczematous or bullous disease | 1 year
Patient survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vivien HEBERT, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- UHRouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No